CLINICAL TRIAL: NCT06552156
Title: FOod Additives on the Mucosal Barrier
Acronym: FOAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: S66308
Record Dates: First submitted 2024-08-01; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Emulsifiers; Dietary emulsifiers; Ultra-processed foods

STUDY DESIGN:
Intervention Model Description: Double Blind, placebo-controlled, randomised controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group assignment was only known by the principal investigator. All other people involved (participants and investigators) were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): The intervention was delivered through three daily brownies. These were 'plain' brownies without any further addition next to the basic ingredients.
  Interventions: Dietary Supplement: Dietary Emulsifier
- Carrageenan (Experimental): Brownies that contained k-CGN (375 mg daily, Modernist Pantry, Eliot, ME, USA)
  Interventions: Dietary Supplement: Dietary Emulsifier
- Carboxymethyl Cellulose (CMC) (Experimental): Brownies that contained carboxymethyl cellulose (2.75 g daily, Modernist Pantry, Eliot, ME, USA)
  Interventions: Dietary Supplement: Dietary Emulsifier
- Polysorbate-80 (P80) (Experimental): Brownies that contained polysorbate-80 (1.350 mg daily, Sigma-Aldrich, Darmstad, Germany)
  Interventions: Dietary Supplement: Dietary Emulsifier
- Soy Lecithin (Experimental): Brownies that contained soy lecithin (3.55 g daily, Modernist Pantry, Eliot, ME, USA)
  Interventions: Dietary Supplement: Dietary Emulsifier
- Native Rice Starch (Experimental): Brownies that contained native rice starch (8.72 g daily, Remy B7, BENEO-Remy N.V., Wijgmaal-Leuven, Belgium)
  Interventions: Dietary Supplement: Dietary Emulsifier

INTERVENTIONS:
Dietary Supplement: Dietary Emulsifier — Intervention was delivered by supplying dietary emulsifiers or placebo through 3 brownies a day that participants had to consume.

SUMMARY:
This is a 6-week pilot study in 60 healthy volunteers to explore (1) the effect of an emulsifier-free diet (2) the effect of three dietary emulsifiers which are believed to detrimentally affect human health, (3) and the effect of two neutral alternatives (native rice starch and soy lecithin), compared to placebo on intestinal permeability and inflammation, systemic inflammation, and the gut microbiota.

DETAILED DESCRIPTION:
This is a 6-week randomized, double-blind placebo-controlled pilot study in 60 healthy volunteers to explore (1) the effect of an emulsifier-free diet (2) the effect of dietary emulsifiers carrageenan, CMC, and Polysorbate-80 (which are believed to detrimentally affect human health), (3) and the effect of neutral alternatives (native rice starch and soy lecithin) on intestinal permeability and inflammation, systemic inflammation, and the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* a BMI between 18.5 - 30 kg/m2
* absence of an eating disorder were required.

Exclusion Criteria:

* pregnancy and lactation
* presence of a chronic disease or any known condition resulting in immunosuppression
* past medical history of any eating disorder
* irritable bowel syndrome
* celiac disease
* IBD or any other chronic intestinal disorders
* prior abdominal surgery other than appendectomy or cholecystectomy
* family history of IBD
* current use of non-steroidal anti-inflammatory drugs (NSAIDs), laxatives, anti-diarrheal medication, anticholinergic medications, narcotics, antacids, proton pump inhibitors (PPIs), or dietary supplements that could not be stopped four weeks before the start of the trial
* antibiotic, prebiotic or probiotic use in the past three months before enrollment
* presence of food allergies or intolerance to the components of the study diet
* experienced diarrhoea withing the two weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Intestinal inflammation | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  Faecal calprotectin measurement using stool samples (in mg/kg)
Intestinal paracellular permeability measurements | Baseline - after the emulsifier-free diet (week 2) - at the end of the trial (week 6)
  Intestinal permeability measurements using the lactulose mannitol urinary excretion ratio (LMR) using urine samples
Intestinal transcellular permeability measurements | Baseline - after the emulsifier-free diet (week 2) - - at the end of the trial (week 6)
  Intestinal transcellular permeability measurements using LPS (lipopolysaccharide)-binding protein (LBP) measurement using blood samples.
Gut microbiome composition | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  Assessment of the gut microbial composition using 16S rRNA sequencing of stool samples.
Gut microbiome metabolism | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  Assessment of the gut microbial metabolism faecal short chain fatty acid (SCFA) measurements from stool samples, including acetic acid, propionic acid, and butyric acid.
Systemic inflammation - inflammatory markers | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  OLINK inflammatory proteomic panel using blood samples
Systemic inflammation - CRP | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  C-reactive protein measurement using blood samples
Metabolic health - lipid profile | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  lipid measurements (including LDL-cholesterol, HDL-cholesterol, total cholesterol and triglycerides) using blood samples
Metabolic health - insulin resistance | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  Insulin measurement using blood samples
Metabolic health - fasting glucose | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  Fasting glucose measurements using blood samples
Metabolic health - cardiometabolic markers | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  OLINK cardiometabolic proteomic panel using blood samples
Body composition analysis | Baseline - after the emulsifier-free diet (week 2) - after 2 weeks of the supplementation and the emulsifier-free diet (week 4) - at the end of the trial (week 6)
  bioelectrical impedance analysis (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: João Sabino, MD, Principal Investigator — Leuven University Hospitals
Locations (1):
- University Hospital of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request

REFERENCES:
- [Derived] Wellens J, Vanderstappen J, Hoekx S, Vissers E, Luppens M, Van Elst L, Lenfant M, Raes J, Derrien M, Verstockt B, Ferrante M, Verbeke K, Matthys C, Vermeire S, Sabino J. Effect of Five Dietary Emulsifiers on Inflammation, Permeability, and the Gut Microbiome: A Placebo-controlled Randomized Trial. Clin Gastroenterol Hepatol. 2025 Aug 13:S1542-3565(25)00698-6. doi: 10.1016/j.cgh.2025.08.005. Online ahead of print. PMID 40816342